CLINICAL TRIAL: NCT05838755
Title: A Multicenter Randomized, Double-blind, Placebo-controlled Phase 2 Study to Evaluate Efficacy, Safety, Tolerability, Pharmacokinetics and Target Engagement of GSK3858279 in Adult Participants With Chronic Diabetic Peripheral Neuropathic Pain (DPNP) /NEPTUNE-17
Brief Title: A Study to Evaluate Efficacy and Safety of GSK3858279 in Diabetic Peripheral Neuropathic Pain
Acronym: NEPTUNE-17
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study met futility criteria at pre-planned interim analysis, showing no clinical efficacy of the investigational drug. Based on the lack of efficacy at the interim data review, the sponsor decided to terminate the study.
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 214221; 2022-502313-28-00 (Other: EU-CT)
Record Dates: First submitted 2023-04-20; First posted 2023-05-03 (Actual); Results first posted 2025-11-21 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Pain
Keywords: Diabetes; Neuropathic pain; Diabetic Peripheral Neuropathic Pain (DPNP); 214221; GSK3858279; Efficacy; Safety; Pharmacokinetics; Tolerability
MeSH Terms: conditions — Pain; Diabetes Mellitus; Neuralgia

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Click here to enter text.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- GSK3858279 60 mg (Experimental): Participants received GSK3858279 SC injection 60 milligram (mg) once per week for 12 weeks.
  Interventions: Drug: GSK3858279
- GSK3858279 360 mg (Experimental): Participants received GSK3858279 SC injection 360 mg once per week for 12 weeks.
  Interventions: Drug: GSK3858279
- Placebo (Placebo Comparator): Participants received matching placebo subcutaneous (SC) injection once per week for 12 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GSK3858279 — GSK3858279 was administered
  Arms: GSK3858279 360 mg; GSK3858279 60 mg
Drug: Placebo — Placebo was administered
  Arms: Placebo

SUMMARY:
This is a multicenter randomized, double-blind, placebo-controlled phase 2 study to evaluate efficacy, safety, tolerability, pharmacokinetics, and target engagement of GSK3858279 in adult participants with chronic Diabetic Peripheral Neuropathic Pain (DPNP). The primary objective of the study is to assess the efficacy of GSK3858279 in participants with DPNP who have been unable to sufficiently manage their pain.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be 18-75 years of age inclusive, at the time of signing the informed consent.
* Type I or Type II diabetes with painful, distal, symmetrical, sensory motor neuropathy attributed to diabetes, of at least 6 months duration.
* A pain score ≥4 and less than or equal to (≤) 9 by the 11-point NRS (0-10) for average daily pain intensity over the past 24 hours at the screening visit.
* Body mass index (BMI) within the range 18-40 kilogram per meter square (kg/m^2) (inclusive)
* Capable of giving signed informed consent.

Exclusion Criteria:

* History or presence of cardiovascular, renal, gastrointestinal, lymphatic disorders which in the opinion of the investigator would interfere with the study procedures and/or assessments.
* Participant has current painful peripheral neuropathy due to a cause other than diabetes (e.g. pernicious anemia, hypothyroidism, post-herpetic neuralgia).
* History of significant allergies to monoclonal antibodies.
* Current enrolment or past participation in a clinical study of an investigational medicinal product intervention within the last 30 days or 5 half-lives (whichever is longer) of signing consent.
* Participants who are unlikely to comply with the protocol (e.g. uncooperative attitude, inability to return for subsequent visits, inability to complete the eDiary daily etc.) and/or otherwise considered by the Investigator to be unlikely to complete the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 147 (Actual)
Dates: Start 2023-09-20 (Actual); Primary Completion 2024-10-14 (Actual); Study Completion 2025-02-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (68):
- United States (18):
  - GSK Investigational Site, Anniston, Alabama
  - GSK Investigational Site, Surprise, Arizona
  - GSK Investigational Site, Cerritos, California
  - GSK Investigational Site, Lomita, California
  - GSK Investigational Site, Largo, Florida
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, West Palm Beach, Florida
  - GSK Investigational Site, Decatur, Georgia
  - GSK Investigational Site, Chicago, Illinois
  - GSK Investigational Site, Waltham, Massachusetts
  - GSK Investigational Site, Williamsville, New York
  - GSK Investigational Site, Huntersville, North Carolina
  - GSK Investigational Site, Lancaster, South Carolina
  - GSK Investigational Site, Cypress, Texas
  - GSK Investigational Site, DeSoto, Texas
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, McAllen, Texas
  - GSK Investigational Site, Bellevue, Washington
- Canada (4):
  - GSK Investigational Site, New Westminster, British Columbia
  - GSK Investigational Site, Vancouver, British Columbia
  - GSK Investigational Site, Winnipeg, Manitoba
  - GSK Investigational Site, Toronto, Ontario
- China (7):
  - GSK Investigational Site, Beijing
  - GSK Investigational Site, Guangzhou
  - GSK Investigational Site, Harbin
  - GSK Investigational Site, Luoyang
  - GSK Investigational Site, Shanghai
  - GSK Investigational Site, Wuhan
  - GSK Investigational Site, Yueyang
- France (2):
  - GSK Investigational Site, Corbeil-Essonnes
  - GSK Investigational Site, Mulhouse
- Germany (4):
  - GSK Investigational Site, Bad Homburg
  - GSK Investigational Site, Mainz
  - GSK Investigational Site, Münster
  - GSK Investigational Site, Wallerfing
- Japan (9):
  - GSK Investigational Site, Chiba
  - GSK Investigational Site, Fukuoka
  - GSK Investigational Site, Gunma
  - GSK Investigational Site, Hokkaido
  - GSK Investigational Site, Ibaraki
  - GSK Investigational Site, Kanagawa
  - GSK Investigational Site, Osaka
  - GSK Investigational Site, Tochigi
  - GSK Investigational Site, Tokyo
- Poland (6):
  - GSK Investigational Site, Częstochowa
  - GSK Investigational Site, Gdynia
  - GSK Investigational Site, Katowice
  - GSK Investigational Site, Skorzewo
  - GSK Investigational Site, Sochaczew
  - GSK Investigational Site, Warsaw
- South Africa (5):
  - GSK Investigational Site, Cape Town
  - GSK Investigational Site, Johannesburg
  - GSK Investigational Site, KwaDukuza
  - GSK Investigational Site, Pretoria
  - GSK Investigational Site, Somerset West
- South Korea (3):
  - GSK Investigational Site, Bucheon-si
  - GSK Investigational Site, Daejeon
  - GSK Investigational Site, Seoul
- Spain (6):
  - GSK Investigational Site, A Coruña
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Málaga
  - GSK Investigational Site, Palma de Mallorca
  - GSK Investigational Site, San SebastiAn de Los Rey
  - GSK Investigational Site, Torrevieja Alicante
- United Kingdom (4):
  - GSK Investigational Site, Cannock
  - GSK Investigational Site, Liverpool
  - GSK Investigational Site, Teesside
  - GSK Investigational Site, West Yorkshire

IPD SHARING:
Plan to Share IPD: No
Qualified researchers may request access to anonymized individual patient-level data (IPD) and related study documents of the eligible studies via the Data Sharing Portal. Details on GSK's data sharing criteria can be found at: https://www.gsk.com/en-gb/innovation/trials/data-transparency/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 147 participants were enrolled in the study, Out of which 144 participants were included in the full analysis set (FAS) population.
Pre-assignment Details: A total of 147 participants were enrolled in the study. Three participants were randomized but did not receive any study drug, hence were excluded from the FAS.
Period: Overall Study
Arm/Group | Placebo | GSK3858279 60 mg | GSK3858279 360 mg
Started (Randomized) | 50 | 48 | 49
Full Analysis Set (Full Analysis Set included all randomized participants who received at least one dose of study intervention.) | 48 | 48 | 48
Completed | 20 | 17 | 17
Not Completed | 30 | 31 | 32
Not completed — Adverse Event | 1 | 0 | 0
Not completed — Lack of Efficacy | 1 | 0 | 1
Not completed — Lost to Follow-up | 0 | 1 | 4
Not completed — Withdrawal by Subject | 0 | 2 | 0
Not completed — Study terminated by sponsor | 26 | 27 | 26
Not completed — Randomized, not treated | 2 | 0 | 1
Not completed — Pregnancy | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: The analysis was performed on the Full Analysis Set (FAS) set that included all randomized participants who received at least one dose of study intervention.
Groups:
- GSK3858279 60 mg: Participants received GSK3858279 SC injection 60 mg once per week for 12 weeks.
- Total: Total of all reporting groups
Arm/Group | Placebo | GSK3858279 60 mg | GSK3858279 360 mg | Total
Number analyzed (Participants) | 48 | 48 | 48 | 144
Age, Continuous [Mean (Standard Deviation); unit: YEARS] | 61.3 (8.59) | 60.1 (10.18) | 60.2 (9.26) | 60.5 (9.32)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 19 | 22 | 62
  Male | 27 | 29 | 26 | 82
Race/Ethnicity, Customized [Number; unit: Participants] — [1] The 'All Other Races' category (American Indian or Alaska Native, Black or African American, Asian, Multiple, Not Reported and Unknown) are combined into one category to maintain participant confidentiality and privacy.
  Participants
    White | 30 | 24 | 25 | 79
    American Indian or Alaska Native | 0 | 2 | 0 | 2
    Asian | 15 | 12 | 14 | 41
    Black or African American | 1 | 8 | 9 | 18
    Mixed race | 1 | 1 | 0 | 2
    Not reported | 0 | 1 | 0 | 1
    Unknown | 1 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Weekly Average of Average Daily Pain Score at Week 12, Assessed on the Numeric Rating Scale (NRS)
Description: The change from baseline (CFB) in the weekly average of the average daily pain score at Week 12 was assessed using Numeric Rating Scale (NRS). Participants recorded their average daily pain response daily using a Brief Pain Inventory Item 5. It is a single item designed for self-reporting average pain score for past 24 hours. Participants were asked to mark their average pain intensity daily, using the NRS, on an 11-point scale (0 = no pain, 10 = worst pain imaginable). The weekly average was computed as weekly average of the average daily scores (range: 0-10), where higher scores indicate more severe pain. A negative CFB indicates pain improvement. Baseline was defined as the average score over the 7 days before dosing (Day -7 to -1). Posterior mean CFB and the 95% credible interval were derived using a Bayesian mixed model repeated measures analysis. The data presented as "Mean" refers to the 'posterior mean' and "95% confidence interval" to '95% credible interval'.
Time Frame: Baseline (Day -7 to Day -1) and Week 12
Population: The analysis was performed on the Full Analysis Set population that included all randomized participants who received at least one dose of study intervention. Number of participants with analyzable outcome (measured outcome used in estimation or imputed outcome based on composite intercurrent event strategy) at the current time point were included in the Overall Number of Participants Analyzed field.
Measure: Mean (95% Confidence Interval); unit: Scores on a Scale
Arm/Group | Placebo | GSK3858279 60 mg | GSK3858279 360 mg
Number analyzed (Participants) | 33 | 32 | 32
Scores on a Scale | -1.85 (-2.44) [-2.44 to -1.28] | -2.50 (-3.09) [-3.09 to -1.91] | -2.07 (-2.67) [-2.67 to -1.48]
Statistical Analysis 1: Comparison: Placebo vs GSK3858279 60 mg; Test type: Other — Analysis performed using a Bayesian mixed model repeated measures adjusting for treatment, week, baseline, region and the treatment by week and baseline by week interactions using vague priors; Posterior Mean Difference = -0.65, 95% CI 2-sided [-1.47 to 0.18] — Posterior mean difference with 95% credible interval is reported using Bayesian mixed model repeated measures analysis
Statistical Analysis 2: Comparison: Placebo vs GSK3858279 360 mg; Test type: Other — [test comment as in outcome 1, analysis 1]; Posterior Mean Difference = -0.22, 95% CI 2-sided [-1.04 to 0.61] — Posterior mean difference with 95% credible interval is reported using Bayesian mixed model repeated measures analysis

2. Secondary Outcome: Number of Participants With Adverse Events (AEs), Serious AE (SAEs) and AEs of Special Interest (AESI)
Description: Adverse events, SAEs, and AESIs were collected. An AE is any untoward medical occurrence in participant, temporally associated with use of study intervention, whether or not considered related to medicinal product. Any untoward event resulting in death, life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, congenital anomaly/birth defect, medically important were categorized as SAE. AESIs of the study drug includes serious and opportunistic infections, tuberculosis (TB), serious hypersensitivity reactions and Injection site reactions.
Time Frame: Up to 27 weeks
Population: This analysis was performed on Safety Set which included all participants who received at least 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | GSK3858279 60 mg | GSK3858279 360 mg
Number analyzed (Participants) | 48 | 48 | 48
Participants
  Any AE | 27 | 23 | 24
  Any SAE | 4 | 2 | 0
  Any AESI | 6 | 4 | 5

3. Secondary Outcome: Number of Participants With Greater Than Or Equal To (>=) Grade 3 Hematological/Clinical Chemistry Abnormalities According to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE)
Description: The laboratory measurements included hematology and clinical chemistry. The parameters evaluated were Eosinophils, Hemoglobin, White blood cell, Lymphocyte count, Neutrophil count and Platelet count, Alanine aminotransferase, Alkaline phosphatase, Aspartate aminotransferase, Blood bilirubin, Hypercalcemia, Hypocalcemia, Cholesterol, Creatine Phosphokinase, Creatinine, Gamma Glutamyl Transferase (GGT), Hypoglycemia, Hyperkalemia, Hypernatremia and Hypertriglyceridemia. Worst case grade (G) increase from baseline grade was evaluated for all the laboratory tests that were gradable by National Cancer Institute Common Terminology Criteria (NCI CTCAE). Data is presented for only those parameters for which participants had worst case >= Grade 3 increase from Baseline.
Time Frame: Up to 27 weeks
Population: This analysis was performed on Safety Set which included all participants who received at least 1 dose of study treatment. Only those participants who were measured and analyzed (i.e., contributed data reported in the table) were included in the Overall Number of Participants Analyzed field. 'Number Analyzed' signifies participants evaluable for specified time points.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | GSK3858279 60 mg | GSK3858279 360 mg
Number analyzed (Participants) | 46 | 46 | 46
Participants
  >= Grade 3 increase in Hematological Abnormalities: number analyzed (Participants) | 45 | 46 | 46
  >= Grade 3 increase in Hematological Abnormalities | 0 | 0 | 0
  Grade3 increase-Clinical Chemistry Abnormality,GGT | 0 | 1 | 0

4. Secondary Outcome: Maximum Concentration (Cmax) of GSK3858279
Description: Blood samples were collected for the determination of serum concentrations of GSK3858279 from which pharmacokinetic (PK) parameters were determined. Cmax was predicted from the population PK model fitted to GSK3859279 serum concentration time data collected at the indicated time points for PK analysis.
Time Frame: Pre-dose, Week 1, Week 4, Week 7, Week 8, Week 11, Week 12, Week 16, Week 20 and Week 27 post dose
Population: This analysis was performed on Pharmacokinetic (PK) set which included all randomized participants in the Safety Population who had at least 1 dose of GSK3858279 and at least 1 non-missing PK assessment (Non-quantifiable [NQ] values were considered as non-missing values). Only those participants with data available at specified time points have been analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram per milliliter (ng/mL)
Arm/Group | GSK3858279 60 mg | GSK3858279 360 mg
Number analyzed (Participants) | 25 | 25
Nanogram per milliliter (ng/mL) | 2943.3 (58) [lower limit 58] | 17125.9 (34) [lower limit 34]

5. Secondary Outcome: Time to Maximum Concentration (Tmax) of GSK3858279
Description: Blood samples were collected for the determination of serum concentrations of GSK3858279 from which PK parameters were determined. Tmax was predicted from the population PK model fitted to GSK3859279 serum concentration time data collected at the indicated time points for PK analysis.
Time Frame: Pre-dose, Week 1, Week 4, Week 7, Week 8, Week 11, Week 12, Week 16, Week 20 and Week 27 post dose
Population: The analysis was performed on Pharmacokinetic (PK) set which included all randomized participants in the Safety Population who had at least 1 dose of GSK3858279 and at least 1 non-missing PK assessment (Non-quantifiable [NQ] values were considered as non-missing values). Only those participants with data available at specified time points have been analyzed.
Measure: Median (Full Range); unit: Day
Arm/Group | GSK3858279 60 mg | GSK3858279 360 mg
Number analyzed (Participants) | 25 | 25
Day | 1.518 (0.64) [0.64 to 2.92] | 1.360 (0.47) [0.47 to 6.32]

6. Secondary Outcome: Trough Concentration at the End of the Dosing Interval (Ctau) of GSK3858279
Description: Blood samples were collected for the determination of serum concentrations of GSK3858279 from which PK parameters were determined. Ctau is defined as the lowest concentration reached by a drug before the next dose is administered. Ctau was predicted from the population PK model fitted to GSK3859279 serum concentration time data collected at the indicated time points for PK analysis.
Time Frame: Pre-dose, Week 1, Week 4, Week 7, Week 8, Week 11, Week 12, Week 16, Week 20 and Week 27 post dose
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram per milliliter (ng/mL)
Arm/Group | GSK3858279 60 mg | GSK3858279 360 mg
Number analyzed (Participants) | 25 | 25
Nanogram per milliliter (ng/mL) | 1910.4 (52) [lower limit 52] | 9543.2 (43) [lower limit 43]

7. Secondary Outcome: Average Concentration Over a Dosing Interval (Cavg) of GSK3858279
Description: Blood samples were collected for the determination of serum concentrations of GSK3858279 from which PK parameters were determined. Cavg is the average concentration over the dosing interval (weekly). Cavg was predicted from the population PK model fitted to GSK3859279 serum concentration time data collected at the indicated time points for PK analysis.
Time Frame: Pre-dose, Week 1, Week 4, Week 7, Week 8, Week 11, Week 12, Week 16, Week 20 and Week 27 post dose
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram per milliliter (ng/mL)
Arm/Group | GSK3858279 60 mg | GSK3858279 360 mg
Number analyzed (Participants) | 25 | 25
Nanogram per milliliter (ng/mL) | 2461.8 (54) [lower limit 54] | 13550.4 (35) [lower limit 35]

8. Secondary Outcome: Area Under the Time-Concentration Curve (AUC) Over the Dosing Interval (AUC[0-Tau]) of GSK3858279
Description: Blood samples were collected for the determination of serum concentrations of GSK3858279 from which PK parameters were determined. AUC(0-tau) was predicted from the population model fitted to GSK3859279 serum concentration time data collected at the indicated time points for PK analysis.
Time Frame: Pre-dose, Week 1, Week 4, Week 7, Week 8, Week 11, Week 12, Week 16, Week 20 and Week 27 post dose
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Day*Nanogram per milliliter (Day*ng/mL)
Arm/Group | GSK3858279 60 mg | GSK3858279 360 mg
Number analyzed (Participants) | 25 | 25
Day*Nanogram per milliliter (Day*ng/mL) | 17232.4 (54) [lower limit 54] | 94852.5 (35) [lower limit 35]

9. Secondary Outcome: Change From Baseline in the Short-Form Mcgill Pain Questionnaire Total Score Over Time
Description: The McGill pain questionnaire Short Form 2 is a 22-item questionnaire total score, which evaluated multi-dimensional pain over time. The questionnaire consists of 22 different descriptors of pain, and each item is rated based on a 0-10 pain intensity scale with 0 indicating no pain and 10 as worst possible pain. The total score was calculated as the mean of all item ratings. Higher scores indicate more severe pain. Baseline is defined as the last assessment prior to the first dose with a non-missing value, including those from unscheduled visits. Posterior mean change from baseline, 95 percent (%) credible interval (CI) was derived using Bayesian mixed model repeated measures. The data presented as 'Mean' refers to 'posterior mean' and '95% confidence interval' refers to '95% credible intervals'.
Time Frame: Baseline (Day1), Week 2, Week 4, Week 8 and Week 12
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: Scores on a Scale
Arm/Group | Placebo | GSK3858279 60 mg | GSK3858279 360 mg
Number analyzed (Participants) | 41 | 40 | 43
Scores on a Scale
  Week 2 | -1.39 [-1.80 to -0.97] | -1.04 [-1.46 to -0.61] | -1.49 [-1.91 to -1.07]
  Week 4: number analyzed (Participants) | 39 | 39 | 37
  Week 4 | -1.77 [-2.25 to -1.29] | -1.36 [-1.86 to -0.87] | -1.44 [-1.95 to -0.94]
  Week 8: number analyzed (Participants) | 37 | 34 | 36
  Week 8 | -1.84 [-2.36 to -1.33] | -1.99 [-2.53 to -1.46] | -1.96 [-2.49 to -1.43]
  Week 12: number analyzed (Participants) | 32 | 28 | 29
  Week 12 | -2.07 [-2.65 to -1.49] | -2.25 [-2.85 to -1.65] | -1.89 [-2.49 to -1.29]

10. Secondary Outcome: Change From Baseline in the Weekly Average of Average Daily Pain Score Over Time, Assessed on the NRS
Description: The change from baseline (CFB) in the weekly average of the average daily pain score at indicated time points was assessed using NRS. Participants recorded their average daily pain response daily using a Brief Pain Inventory Item 5. It is a single item designed for self-reporting average pain score for past 24 hours. Participants were asked to mark their average pain intensity daily, using the NRS, on an 11-point scale (0 = no pain, 10 = worst pain imaginable). The weekly average was computed as weekly average of the average daily scores (range: 0-10), where higher scores indicate more severe pain. A negative CFB indicates pain improvement. Baseline was defined as the average score over the 7 days before dosing (Day - 7 to -1). Posterior mean CFB and the 95% credible interval were derived using a Bayesian mixed model repeated measures analysis. The data presented as 'Mean' refers to the 'posterior mean' and '95% confidence interval' to the '95% credible interval'.
Time Frame: Baseline (Day -7 to Day -1), Week 1, Week 2, Week 3, Week 4, Week 5, Week 6, Week 7, Week 8, Week 9, Week 10, Week 11 and Week 12
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: Scores on a Scale
Arm/Group | Placebo | GSK3858279 60 mg | GSK3858279 360 mg
Number analyzed (Participants) | 48 | 48 | 48
Scores on a Scale
  Week 1 | -0.47 [-0.76 to -0.17] | -0.57 [-0.87 to -0.27] | -0.68 [-0.98 to -0.38]
  Week 2: number analyzed (Participants) | 46 | 46 | 45
  Week 2 | -0.71 [-1.10 to -0.32] | -0.95 [-1.34 to -0.55] | -1.16 [-1.55 to -0.76]
  Week 3: number analyzed (Participants) | 44 | 45 | 44
  Week 3 | -0.94 [-1.37 to -0.50] | -1.24 [-1.68 to -0.80] | -1.50 [-1.94 to -1.06]
  Week 4: number analyzed (Participants) | 41 | 42 | 39
  Week 4 | -1.34 [-1.81 to -0.87] | -1.42 [-1.90 to -0.94] | -1.60 [-2.08 to -1.11]
  Week 5: number analyzed (Participants) | 40 | 40 | 39
  Week 5 | -1.54 [-2.09 to -1.00] | -1.60 [-2.16 to -1.04] | -1.74 [-2.30 to -1.18]
  Week 6: number analyzed (Participants) | 39 | 40 | 39
  Week 6 | -1.59 [-2.12 to -1.07] | -1.71 [-2.24 to -1.18] | -1.73 [-2.26 to -1.20]
  Week 7: number analyzed (Participants) | 38 | 39 | 39
  Week 7 | -1.63 [-2.18 to -1.09] | -1.91 [-2.46 to -1.35] | -1.94 [-2.50 to -1.38]
  Week 8: number analyzed (Participants) | 37 | 36 | 37
  Week 8 | -1.72 [-2.27 to -1.18] | -2.10 [-2.66 to -1.54] | -1.99 [-2.55 to -1.43]
  Week 9: number analyzed (Participants) | 37 | 37 | 37
  Week 9 | -1.71 [-2.25 to -1.18] | -2.13 [-2.67 to -1.59] | -1.94 [-2.49 to -1.40]
  Week 10: number analyzed (Participants) | 36 | 35 | 34
  Week 10 | -1.76 [-2.30 to -1.22] | -2.31 [-2.86 to -1.76] | -2.01 [-2.56 to -1.45]
  Week 11: number analyzed (Participants) | 35 | 33 | 33
  Week 11 | -1.88 [-2.44 to -1.32] | -2.40 [-2.98 to -1.83] | -2.12 [-2.70 to -1.55]
  Week 12: number analyzed (Participants) | 33 | 32 | 32
  Week 12 | -1.85 [-2.44 to -1.28] | -2.50 [-3.09 to -1.91] | -2.07 [-2.67 to -1.48]

11. Secondary Outcome: Proportion of Participants With Greater Than or Equal To (>=) 30 Percentage (%) Reduction From Baseline in the Weekly Average of Average Daily Pain Intensity at Week 12, Assessed on the NRS
Description: The proportion of participants who achieved >=30 percentage reduction from Baseline (responders) in the weekly average of the average daily pain score at Week 12 as measured by NRS is reported. Participants were instructed to assess their average daily pain daily, and to record the response in a Brief Pain Inventory item 5. It is a single item designed to capture information on the self- reported average pain score over the past 24 hours. Participants were asked to mark their pain- intensity daily, using the NRS, on an 11- point scale (0-10), with 0 = no pain, and 10 = worst pain imaginable. The weekly average was computed as weekly average of the average daily scores (range: 0-10), where higher scores indicate more severe pain. The data is presented for proportion of responders where 'Mean' refers to 'posterior mean proportion' and '95% confidence interval' refers to '95% credible interval'.
Time Frame: At Week 12
Population: The analysis was performed on the Full Analysis Set (FAS) set that included all randomized participants who received at least one dose of study intervention. Only those participants who were measured and analyzed (i.e., contributed data reported in the table) were included in the Overall Number of Participants Analyzed field. 'Number Analyzed' signifies participants evaluable for specified time points.
Measure: Mean (95% Confidence Interval); unit: Proportion of participants
Arm/Group | Placebo | GSK3858279 60 mg | GSK3858279 360 mg
Number analyzed (Participants) | 33 | 32 | 32
Proportion of participants | 0.50 (0.38) [0.38 to 0.62] | 0.64 (0.52) [0.52 to 0.75] | 0.55 (0.43) [0.43 to 0.67]

12. Secondary Outcome: Proportion of Participants With Greater Than or Equal To >= 50 % Reduction From Baseline in the Weekly Average of Average Daily Pain Score at Week 12, Assessed on the NRS
Description: The proportion of participants who achieved >=50 percentage reduction from Baseline (responders) in the weekly average of the average daily pain score at Week 12 as measured by NRS is reported. Participants were instructed to assess their average daily pain daily, and to record the response in a Brief Pain Inventory item 5. It is a single item designed to capture information on the self- reported average pain score over the past 24 hours. Participants were asked to mark their pain- intensity daily, using the NRS, on an 11- point scale (0-10), with 0 = no pain, and 10 = worst pain imaginable. The weekly average was computed as weekly average of the average daily scores (range: 0-10), where higher scores indicate more severe pain. The data is presented for proportion of responders where 'Mean' refers to 'posterior mean proportion' and '95% confidence interval' refers to '95% credible interval'.
Time Frame: At Week 12
Population: as for outcome 11
Measure: Mean (95% Confidence Interval); unit: Proportion of participants
Arm/Group | Placebo | GSK3858279 60 mg | GSK3858279 360 mg
Number analyzed (Participants) | 33 | 32 | 32
Proportion of participants | 0.28 (0.19) [0.19 to 0.39] | 0.40 (0.29) [0.29 to 0.52] | 0.32 (0.22) [0.22 to 0.44]

ADVERSE EVENTS:
Time Frame: All-cause mortality, Serious Adverse Events (SAEs) and non-Serious Adverse Events (non-SAEs) were collected from the start of the study intervention (Day 1) until follow up of week 27.
Description: Safety set included all randomized participants who took at least 1 dose of study intervention. Participants were analyzed according to the treatment they actually received.
Groups:
- Placebo: Participants received placebo SC injection once per week for 12 weeks.
- GSK3858279 60 Milligram (mg) Weekly: Participants received GSK3858279 subcutaneous (SC) injection 60 mg once per week for 12 weeks.
- GSK3858279 360 mg Weekly: Participants received GSK3858279 SC injection 360 mg once per week for 12 weeks.
Arm/Group | Placebo | GSK3858279 60 Milligram (mg) Weekly | GSK3858279 360 mg Weekly
All-Cause Mortality (participants affected / at risk) | 0/48 | 0/48 | 0/48
Serious Adverse Events (participants affected / at risk) | 4/48 | 2/48 | 0/48
Other Adverse Events (participants affected / at risk) | 11/48 | 9/48 | 10/48
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=48) | GSK3858279 60 Milligram (mg) Weekly (N=48) | GSK3858279 360 mg Weekly (N=48)
Angina unstable (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cat scratch disease (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Hemianopia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=48) | GSK3858279 60 Milligram (mg) Weekly (N=48) | GSK3858279 360 mg Weekly (N=48)
Injection site haemorrhage (General disorders) | 0 (0) | 0 (0) | 3 (6)
Bronchitis (Infections and infestations) | 1 (1) | 1 (1) | 3 (3)
COVID-19 (Infections and infestations) | 0 (0) | 4 (4) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 3 (3) | 2 (2) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (4) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (7) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 3 (3)
Headache (Nervous system disorders) | 5 (7) | 2 (2) | 2 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2024-03-26): https://cdn.clinicaltrials.gov/large-docs/55/NCT05838755/Prot_000.pdf
  • Statistical Analysis Plan (2025-01-30): https://cdn.clinicaltrials.gov/large-docs/55/NCT05838755/SAP_001.pdf